CLINICAL TRIAL: NCT03055273
Title: SOCIABLE Seniors Optimizing Community Integration to Advance Better Living With ESRD
Acronym: SOCIABLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Roybal Center (Unknown); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NA00097283; P30AG048773 (NIH)
Record Dates: First submitted 2016-08-31; First posted 2017-02-16 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: ESRD; Social Behavior; Physical Disability
MeSH Terms: conditions — Kidney Failure, Chronic; Social Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SOCIABLE IMMEDIATE (Experimental): Receive services now
  Interventions: Behavioral: SOCIABLE
- SOCIABLE wait list (Active Comparator): Receive services four months post-enrollment
  Interventions: Behavioral: SOCIABLE

INTERVENTIONS:
Behavioral: SOCIABLE — SOCIABLE services involve a nurse, and occupational therapist and a handyman to support function among older adults with end stage renal disease. There is particular emphasis on supporting the social function and the physical and everyday living function.

SUMMARY:
This research is being done to find out the best ways to help people with end stage kidney disease take care of their daily lives and improve their social functioning.

Investigators want to learn whether services in the Community Aging in Place, Advancing Better Living for Elders (CAPABLE) study such as help with medications, muscle strengthening, balance training, pain management, changes to houses and improved social support can be tailored to fit the needs of older adults with kidney disease to help improve their ability to balance, walk, and take care of themselves.

People aged 60 years and older who have end stage kidney disease and have been receiving dialyses for at least 6 months, may join.

DETAILED DESCRIPTION:
Questionnaires:

Participants will be asked to answer questions about:

* social support and social functioning
* pain and depression
* physical function

Study intervention:

Participants will be randomly assigned (by chance, like the flip of a coin) to one of two groups: participant either will receive SOCIABLE (Seniors Optimizing Community Integration to Advance Better Living with ESRD) services now, or will receive the same services in six months from now. Participants have a 50:50 chance of getting into each group

SOCIABLE services involve receiving visits with a nurse interviewer. Participants will decide how you want to improve your social function and social support.

Participants will also receive:

* a group of services called CAPABLE which include home visits from a nurse (RN) and an occupational therapist (OT) and a handyman for repairs if you need them and
* help with improving social support

All participants will receive 10 home visits (6 OT, 4 RN) plus minor home repairs and assistive devices over a 4 month period of time.

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older
* End Stage Renal Disease on In-Center Hemodialysis for at least 6 months
* Functional limitations (difficulty in at least one of the following: bathing, dressing, walking across a room, grooming, getting on or off the toilet, getting on or off the bed);
* Low socioeconomic status (less than high School education, or household income <$25,000/year)
* Signed informed consent

Exclusion Criteria:

* Inability to understand the informed consent process and give consent via signed written consent form

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Katz ADL | baseline
  Questionnaire about Activities of Daily Living such as bathing, dressing, walking, grooming and how difficult each one is to do. 8 questions and they range from 0, meaning they have no difficulty to 2 which means they can not do it even with help.
Katz ADL | 4 months post intervention
  Questionnaire about Activities of Daily Living such as bathing, dressing, walking, grooming and how difficult each one is to do. 8 questions and they range from 0, meaning they have no difficulty to 2 which means they can not do it even with help.
Katz ADL | 8 months post intervention
  Questionnaire about Activities of Daily Living such as bathing, dressing, walking, grooming and how difficult each one is to do. 8 questions and they range from 0, meaning they have no difficulty to 2 which means they can not do it even with help.

SECONDARY OUTCOMES:
Lawton Instrumental Activities of Daily Living (IADL) measure | Baseline
  This questionnaire measures participants' abilities to do Instrumental Activities of Daily Living such as shopping, light housekeeping, and managing finances. The scale ranges from 0 meaning they have no difficulty to 2 which means they can't do it even if they have help
Lawton Instrumental Activities of Daily Living (IADL) measure | 4 months
  This questionnaire measures participants' abilities to do Instrumental Activities of Daily Living such as shopping, light housekeeping, and managing finances. The scale ranges from 0 meaning they have no difficulty to 2 which means they can't do it even if they have help
Lawton Instrumental Activities of Daily Living (IADL) measure | 8 months
  This questionnaire measures participants' abilities to do Instrumental Activities of Daily Living such as shopping, light housekeeping, and managing finances. The scale ranges from 0 meaning they have no difficulty to 2 which means they can't do it even if they have help

CONTACTS AND LOCATIONS:
Overall Officials: Deidra Crews, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided